CLINICAL TRIAL: NCT04677140
Title: Hip Related Functional Limitations in Individuals With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Çelik, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/694
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Scoliosis Idiopathic
Keywords: scoliosis; hip; jaw; adolescent idiopathic scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experiment group: By a specialist physician with existing anteroposterior and lateral radiographs have been diagnosed with adolescent idiopathic scoliosis

SUMMARY:
The aim of this study is to examine the functional parameters of hip and jaw in terms of scoliosis degree and scoliosis pattern in individuals with idiopathic scoliosis.

DETAILED DESCRIPTION:
In this study investigators will examine the hip functional parameters and jaw functional parameters separately.

In hip study hip functional parameters will be evaluated for determining the correlation between scoliosis degree/pattern and hip functions.

In jaw study jaw functional parameters will be evaluated for determining the correlation between scoliosis degree/pattern and hip functions.

ELIGIBILITY:
Inclusion Criteria: (for all hip and jaw evaluation)

* Having been diagnosed with adolescent idiopathic scoliosis by a specialist physician with existing anterior-posterior and lateral lateral radiographs,
* Primary curvature over 10 degrees in the coronal plane according to the Cobb method,
* Being literate,
* To cooperate in answering and implementing evaluation scales,
* Children with written consent from their parents and themselves will be included.

Exclusion Criteria: (for hip evaluation)

* Having any systemic illness,
* Spinal surgery history,
* Presence of any acute or chronic disease other than scoliosis,
* Inadequate quality to examine the measurement parameters of the current vertebral radiography,
* Use of musical instruments,
* Long-term and professional sports.

Exclusion Criteria: (for jaw evaluation)

* Having any systemic illness,
* Spinal surgery history,
* Presence of any acute or chronic disease other than scoliosis,
* Aesthetics or any injection intervention in the face and neck area,
* Spinal surgery history,
* Orthodontic treatment,
* Use of musical instruments,
* Long-term and professional sports.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Our study will include cases who applied to Hacettepe University, Faculty of Physical Medicine and Rehabilitation with a diagnosis of scoliosis, had anterior-posterior and lateral radiographs, accepted to participate in the study on a voluntary basis, were literate and cooperated in completing the scales. In cases under the age of 18, the evaluation will be started by obtaining additional family consent.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
single leg squat test (SLS) | Baseline
  single leg squat test will be evaluated for each patient (min:0, max:3)

SECONDARY OUTCOMES:
Y balance test (YBT) | Baseline
  Y balance test will be evaluated (cm)

OTHER OUTCOMES:
Hip ROM (range of motion) | Baseline
  Hip ROM (range of motion) will be evaluated with goniometer (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Yağcı, Study Director — associate professor
Locations (1):
- Hacettepe University Physical Therapy and Rehabilitation Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choudhry MN, Ahmad Z, Verma R. Adolescent Idiopathic Scoliosis. Open Orthop J. 2016 May 30;10:143-54. doi: 10.2174/1874325001610010143. eCollection 2016. PMID 27347243